CLINICAL TRIAL: NCT05191004
Title: Randomized, Non-Comparative Phase 1/2 Study of NUV-422 in Combination With Fulvestrant in Patients With Hormone Receptor-Positive Human Epidermal Growth Factor Receptor 2-Negative (HR+HER2-) Advanced Breast Cancer (aBC)
Brief Title: Study of NUV-422 in Combination With Fulvestrant in Patients With HR+HER2- aBC
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NUV-422-03
Record Dates: First submitted 2021-12-22; First posted 2022-01-13 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer; Breast Cancer; Breast Carcinoma; Cancer of the Breast; Cancer of Breast; Malignant Tumor of Breast; Breast Tumor
Keywords: Phase 1; Phase 2; metastatic breast cancer; advanced breast cancer; hormone receptor positive; HR+; human epidermal growth factor receptor 2 negative; HER2-; HR+ HER2-; estrogen receptor positive; ER+; NUV-422; fulvestrant; CDK; CDK inhibition; CDK2/4/6
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: Sequential assignment or parallel assignment will be applied (in both Phase 1 and Phase 2), depending on the stage of the study at the time of a patient's enrollment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1b Dose Escalation (Experimental): NUV-422 will be administered orally at escalating dose levels in combination with fulvestrant until the recommended Phase 2 combination dose (RP2cD) is determined.
  500 mg fulvestrant will be administered IM on Days 1 and 15 of Cycle 1 and Day 1 of every cycle thereafter.
  Interventions: Drug: NUV-422; Drug: Fulvestrant
- Phase 2 NUV-422 + fulvestrant (Experimental): NUV-422 will be administered orally at the RP2cD in combination with fulvestrant.
  500 mg fulvestrant will be administered IM on Days 1 and 15 of Cycle 1 and Day 1 of every cycle thereafter.
  Interventions: Drug: NUV-422; Drug: Fulvestrant
- Phase 2 NUV-422 monotherapy (Experimental): NUV-422 will be administered orally at the RP2cD.
  Interventions: Drug: NUV-422
- Phase 2 fulvestrant monotherapy (Experimental): 500 mg fulvestrant will be administered IM on Days 1 and 15 of Cycle 1 and Day 1 of every cycle thereafter.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: NUV-422 — NUV-422 is an investigational drug for oral dosing.
  Arms: Phase 1b Dose Escalation; Phase 2 NUV-422 + fulvestrant; Phase 2 NUV-422 monotherapy
Drug: Fulvestrant — Fulvestrant
  Other Names: Faslodex
  Arms: Phase 1b Dose Escalation; Phase 2 NUV-422 + fulvestrant; Phase 2 fulvestrant monotherapy

SUMMARY:
NUV-422-03 is a randomized, non-comparative Phase 1/2 dose escalation and expansion study designed to evaluate the safety and efficacy of NUV-422 in combination with fulvestrant relative to NUV-422 monotherapy and fulvestrant monotherapy. The study population is comprised of adults with HR+HER2- aBC. Patients will self-administer NUV-422 orally in 28-day cycles and receive 500 mg fulvestrant intramuscularly (IM) on Days 1 and 15 of Cycle 1 and Day 1 of every cycle thereafter. Patients will be treated until disease progression, toxicity, withdrawal of consent, or termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with diagnosis of locally advanced inoperable or metastatic HR+HER2- breast cancer
2. Evidence of disease progression on immediate prior therapy as determined by the Investigator per standard criteria
3. Patients must have received standard of care treatments for their breast cancer and be eligible to receive fulvestrant

   * Prior standard of care treatments must include treatment with hormonal therapy in combination with an approved CDK4/6 inhibitor
4. Patients must have endocrine-resistant disease
5. Have no known active or symptomatic central nervous system (CNS) disease
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1
7. Life expectancy of > 6 months
8. Eligible to receive fulvestrant
9. Adequate bone marrow and organ function

Exclusion Criteria:

1. Have received chemotherapy, hormonal therapy (with the exception of ongoing LHRH analogs in male patients and premenopausal women), radiation, or biological anti-cancer therapy within 14 days prior to the first dose of NUV-422 and fulvestrant
2. Received treatment with an investigational agent for any indication within 14 days for non-myelosuppressive agent or 21 days (of < 5 half-lives) for myelosuppressive agent prior to first dose of NUV-422 and fulvestrant
3. Moderate liver impairment which would require a reduced dose of fulvestrant
4. Requires medications that are known to be strong inducers and/or inhibitors of CYP3A4/5 enzymes

   * For Phase 1b only: requires medications that are known to be moderate inducers and/or inhibitors of CYP3A4/5 enzymes
5. Known allergy or hypersensitivity to fulvestrant
6. For Phase 2 only: prior therapy with fulvestrant and/or investigational ER targeted agent
7. Females who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1b Dose Escalation: Safety and tolerability of NUV-422 in combination with fulvestrant to determine the recommended Phase 2 combination dose (RP2cD) | During the DLT period (28 days)
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), dose-limiting toxicities (DLTs), and laboratory abnormalities
Phase 2 Dose Expansion: Objective Response Rate (ORR) | Every 8 weeks through study treatment, an average of 6 months
  ORR per standard criteria

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Compassionate Cancer Care Research Inc., Fountain Valley, California
  - Gabrail Cancer Center Research, Canton, Ohio
  - Pennsylvania Cancer Specialists and Research Institute, Gettysburg, Pennsylvania
  - NEXT Virginia, Fairfax, Virginia